CLINICAL TRIAL: NCT02386176
Title: The Assessment of the Role of Automated Breast Ultrasound (ABUS) in Screening Women With Dense Breasts for Early Detection of Breast Cancer
Brief Title: Assessment of Automated Breast Ultrasound
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Denise Chough, MD, Associate Professor, University of Pittsburgh
Other Study IDs: PRO14110472
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators are interested in assessing the value of and comparing the use of automated breast ultrasound (ABUS) (either as a primary screening approach or as a supplementary procedure) with digital breast tomosynthesis (DBT). The purpose of this project is to perform a preliminary prospective study on women who are most likely to benefit from the use of ABUS and/or DBT (or a combination of both) in the screening environment.

DETAILED DESCRIPTION:
1. After appropriate training and certification of technologists and Mammography Quality Standards Act (MQSA) qualifications of the participating radiologists, the investigators will recruit sequentially approximately 600 women known to have a defined region of highly dense tissue or with known heterogeneously dense and/or primarily dense breast tissue (from a prior mammogram) who are scheduled to undergo routine mammography screening that includes a DBT examination.
2. Consenting women will undergo a DBT examination as part of their routine clinical exam and an ABUS examination as a part of the experiment. All examinations will be performed by certified technologists in the performance of each of the procedures in question (DBT or ABUS).
3. DBT, ABUS, and a combination of both, will be independently reviewed and interpreted (Breast Imaging, Reporting and Data System rated) by experienced and specifically trained, MQSA qualified radiologists in a cross balanced (cases by mode and by reader) study design.
4. Using the results of the interpretations in a slightly modified "LOGICAL OR" mode, namely the highest rating determines the recommendation/need for follow up, the investigators will perform imaging based diagnostic work ups as needed (i.e., resulting from the "arbitration step"). All diagnostic follow up studies, as needed, will not be a part of the study protocol, with the exception of acquiring diagnostic outcome measures from medical records.
5. The investigators will compare rates of false positives as a result of interpreting DBT vs. ABUS vs. a combination of both, including recall for additional testing, short-interval follow-up rates and biopsy rates. The sample in this preliminary study is too small to assess positive predictive values (PPVs), so the investigators will focus here on negative predictive values (NPVs). For marginal value assessment when utilizing both modalities, the investigators will also assess the type of abnormalities detected by each modality, assuming that a larger study will be required to assess cancer detection rates (by type etc.).

ELIGIBILITY:
Inclusion Criteria:

* 40 to 75 years of age with a
* defined region of extremely dense breast tissue or heterogeneously dense or extremely dense parenchyma by prior digital mammography report (i.e., "dense breasts")
* presenting for routine annual mammography with digital breast tomosynthesis.

Exclusion Criteria:

* Known to be at high risk for breast cancer due to known or suspected pathologic breast cancer susceptibility gene (BRCA) (i.e. first-degree relative with known mutation) or prior chest radiation therapy before age 30;
* No mammogram within the prior 3 years;
* Signs or symptoms of breast disease including lump, bloody or spontaneous clear nipple discharge, eczema of the nipple;
* Pregnancy at the time of screening by self report or lactation within the prior 6 months;
* Breast implants, as assessment of breast density may be problematic;
* Recent prior breast surgery or breast biopsy or cyst aspiration within the prior 12 months;
* Had prior screening with DBT and not a hand held ABUS, or had prior screening with ABUS and not DBT.
* Prior malignancy other than: Breast cancer at least one year earlier (12 full months have elapsed since the last treatment surgery) with no known distant metastases and no known residual tumor, or Basal or squamous cell skin cancer or in situ cervical cancer, or Other cancer for which the patient has been disease free for ≥ 5 years, with no recurrence of cancer in the last five years and no residual disease detected in the last five years
* Unwilling or unable to provide consent.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women aged 40 to 75 years of age with a defined region of extremely dense breast tissue or heterogeneously dense or extremely dense parenchyma by prior digital mammography report (i.e., "dense breasts"), presenting for routine annual mammography with digital breast tomosynthesis.
Sampling Method: Non-Probability Sample
Enrollment: 598 (Actual)
Dates: Start 2015-08; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
false positive rates | from the date interpretation until the date routine follow-up, biopsy results, or pathology results, whichever comes first, up to 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Denise M Chough, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States